CLINICAL TRIAL: NCT04970602
Title: The Effect of Early Use of Methylene Blue on Hemodynamics in Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20210621
Record Dates: First submitted 2021-06-29; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Septic Shock
Keywords: septic shock; methylene blue; vasopressor; refractory shock
MeSH Terms: conditions — Shock, Septic; Shock | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB group (Experimental): This group will be given 2mg/kg methylene blue infusion within 20 minutes, 2 hours later followed by 0.5mg/kg/h for 4 hours.
  Interventions: Drug: Methylene Blue
- control group (No Intervention): This group will be given conventional vasopressors, except methylene blue, based on the attending doctor's decision.

INTERVENTIONS:
Drug: Methylene Blue — Once the patient meets inclusion criterial, the interventional group will receive 2mg/kg methylene blue infusion within 20min, followed by 0.5mg/kg/h for 4 hours.
  Arms: MB group

SUMMARY:
This study will include patients requiring high dose of norepinephrine (NA) to maintain blood pressure after fluid resuscitation. The patients will be randomized into two groups, the study protocol is early combined application of methylene blue. The primary outcome is Sequential Organ Failure Assessment (SOFA) score 72 hours after admission. Second outcome includes duration of shock, length of intensive care unit (ICU) hospitalization and so on. To explore the underlying mechanism, the changes of sublingual microcirculation before and after vasopressor combination will be collected, also is the global longitudinal strain of left ventricle.

DETAILED DESCRIPTION:
Background: Decreased vascular tone is one of the main mechanisms leading to septic shock. The guidelines recommend NA as the first-line vasopressor. The benefits of early combination with other vasopressors are not yet known.

Methods:

1. Patients: Septic shock patients in need of high dose of NA (≥0.5ug/kg.min maintaining more than 2 hours) to maintain blood pressure after fluid resuscitation.
2. Intervention: The patients will be randomized into two groups. The study group will receive 2mg/kg methylene blue infusion with 15 minutes, 2 hours laters followed by 0.5mg/kg/h for 4 hours. The control group received conventional treatments, the attending physicians decide the protocol of vasopressors. The data including patients' characters, duration of shock and hospitalization, duration of mechanical ventilation, cumulative dose of vasopressors will be collected. Before and 6h after meeting the inclusion standard, sublingual microcirculation and automated function imaging of myocardium will be performed.
3. Outcome: The primary outcome is SOFA score 72 hours after admission. Second outcome includes duration of shock, length of ICU hospitalization and so on. the changes of sublingual microcirculation will be collected, also is the global longitudinal strain of left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock, receive 0.5 ug/kg/min NA to maintain blood pressure for more than 2 hours after fluid resuscitation.

Exclusion Criteria:

* Pregnant women
* Without internal jugular vein or subclavian vein catheterization
* Child-Pugh grade C with liver cirrhosis
* Severe chronic obstructive pulmonary disease (severe acidosis caused by type II respiratory failure, PaCO2 ≥60mmHg and PH<7.2 )
* End-stage of malignant tumors
* Glucose-6-phosphate dehydrogenase (G6PD enzyme) deficiency
* Positive end-respiratory pressure (PEEP) >10mmHg, the oxygenation index <150mmHg under mechanical ventilation
* Definitive pulmonary hypertension or chronic pulmonary heart disease.
* Oral use of 5-hydroxytryptamine in recent 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
SOFA score | 72 hours
  72 hours after inclusion

SECONDARY OUTCOMES:
duration of shock | 2 hours
  the duration between diagnosis and relief of septic shock, the latter is defined by stable blood pressure without any vasopressor for 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Xiangya Hospital, Central South University, Principal Investigator — Department of Critical Care Medicine, Xiangya Hospital, Central South University
Locations (1):
- Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, objective data could be shared when required.
Supporting Information: Study Protocol, CSR
Time Frame: Within 1 year after completion of the study.
Access Criteria: Just for academic requirement.